CLINICAL TRIAL: NCT05802979
Title: Analgesic Efficacy of Ketamine Versus Neostigmine as Adjuvants to Bupivacaine During Ultrasound-guided Serratus Anterior Plane Block in Modified Radical Mastectomy
Brief Title: Ketamine Versus Neostigmine as Adjuvants to Bupivacaine During Ultrasound-guided Serratus Anterior Block
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Aya Hisham, Lecturer of Anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FMASU MD 209/2022
Record Dates: First submitted 2023-03-26; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: Post Operative Pain
Keywords: mastectomy; postoperative pain; serratus anterior block; adjuvants
MeSH Terms: conditions — Pain, Postoperative | interventions — Adjuvants, Anesthesia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- group 1 (Active Comparator): consists of patients receiving Serratus anterior plane block using Bupivacaine + Ketamine.
  Interventions: Drug: Adjuvants, Anesthesia
- group 2 (Active Comparator): consists of patients receiving Serratus anterior plane block using Bupivacaine + neostigmine.
  Interventions: Drug: Adjuvants, Anesthesia
- group 3 (Placebo Comparator): consists of patients receiving Serratus anterior plane block using Bupivacaine + normal saline.
  Interventions: Drug: Adjuvants, Anesthesia

INTERVENTIONS:
Drug: Adjuvants, Anesthesia — testing the effect of adding ketamine versus neostigmine to the analgesic efficacy of serratus anterior plane block in modified radical mastectomy surgeries

SUMMARY:
This study is designed to investigate the analgesic efficacy of ketamine compared to neostigmine as adjuvants to LA in ultrasound guided Serratus Anterior Plane Block (SAPB) in patients undergoing Modified Radical Mastectomy. We hypothesize that adding either neostigmine or ketamine to bupivacaine in ultrasound guided SAPB would increase the total analgesic duration and decrease the total 24 hr postoperative Nalbuphine consumption compared to SAPB with bupivacaine only. The first 24 hr of postoperative Nalbuphine consumption is set as the primary outcome. The time of the first request of analgesia, pain score, side effects of drugs and patient hemodynamics are set as the secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* ASA II patients, BMI< 35Kg/m2

Exclusion Criteria:

* refusal of participation, ASA III or above, history of allergy to the study drugs, BMI> 35kg/m2, coagulation disorders, psychiatric illnesses that may interfere with pain evaluation, epileptic patients, patients with tachy or brady arrthymias, patients with increased intracranial tension

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — biologically female patients undergoing mastectomy for breast cancer
Enrollment: 80 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
analgsic consumption | first 24 hours postoperative
  total amount of consumed nalbuphine

SECONDARY OUTCOMES:
time to rescue analgesia | first 24 hours postoperative
  first time to request rescue analgesia
pain scores | first 24 hours postoperative
  pain scores measured by numerical pain score chart

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed S Abd El Aziz, M.D., Study Director — AinShams University
Locations (1):
- AinShams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdelhamid BM, Samy S, Abdalla A, Saad A, Ollaek M, Ahmed A. Ketamine versus neostigmine as adjuvants to bupivacaine during ultrasound-guided serratus anterior plane block in modified radical mastectomy. A randomized controlled trial. Egyptian Journal of Anaesthesia. 2021; 37(1):356-363.
- [Background] Elbahrawy K, El-Deeb A. The effects of adding neostigmine to supraclavicular brachial plexus block for postoperative analgesia in chronic renal failure patients: a prospective randomized double-blinded study. Research and Opinion in Anesthesia and Intensive Care. 2016; 3(1):36-41. Omar AM, Mansour MA, Abdelwahab HH, Aboushanab OH
- [Background] Pandey V, Mohindra BK, Sodhi GS. Comparative evaluation of different doses of intrathecal neostigmine as an adjuvant to bupivacaine for postoperative analgesia. Anesth Essays Res. 2016 Sep-Dec;10(3):538-545. doi: 10.4103/0259-1162.180779. PMID 27746548
- [Background] Rashwan DAEK, Mohammed AR, Kasem Rashwan SA, Abd El Basset AS, Nafady HA. Efficacy of Serratus Anterior Plane Block Using Bupivacaine/ Magnesium Sulfate Versus Bupivacaine/ Nalbuphine for Mastectomy: A Randomized, Double-Blinded Comparative Study. Anesth Pain Med. 2020 Jun 22;10(3):e103141. doi: 10.5812/aapm.103141. eCollection 2020 Jun. PMID 32944562